CLINICAL TRIAL: NCT06828120
Title: A Randomized, Safety and Efficacy Study of Taneasy 600mg Granules and Fluimucil 600mg Granules in COPD Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bun Yao Biotechnology Co., Ltd (Industry)
Collaborators: Clinny biotech limited (Unknown); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCQ230209TP
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taneasy 600mg granules (Experimental): Dose： 600 mg/time. Use ：two times per day.
- Fluimucil 600mg granules (Active Comparator): Dose： 600 mg/time. Use ：two times per day

INTERVENTIONS:
Drug: Taneasy 600mg granules — Treatment of respiratory affections characterized by thick and viscous hypersecretion due to acute bronchitis,chronic bronchitis and its exacerbation, plumonary emphysema,mucoviscidosis and bronchiectasis.
Drug: Fluimucil 600mg granules — Treatment of respiratory affections characterized by thick and viscous hypersecretion due to acute bronchitis,chronic bronchitis and its exacerbation, plumonary emphysema,mucoviscidosis and bronchiectasis.

SUMMARY:
To evaluate the safety and efficacy of Taneasy 600mg granules and Fluimucil 600mg granules administered twice daily for 14 days in treatment of COPD Disease.

DETAILED DESCRIPTION:
The study will enroll 40~60 patients and complete 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged older than 20~75 years old.
* Able to sign informed consent prior to the study.
* The appearance of sputum and the difficulty of expectoration are both at level 2 or above.

Exclusion Criteria:

* Subjects with known hypersensitivity to Acetylcysteine preparations.
* Subjects with other serious medical diseases that are judged by the attending physician to affect the evaluation results (such as: tuberculosis, pneumonia, bronchial asthma, bronchiectasis, cor pulmonale, lung cancer, acute myocardial infarction, acute hepatitis, renal failure, etc.)
* Pregnancy or breast-feeding woman.
* Female subjects or their sexual partners do not use contraception during the trial.
* Joining any drug clinical trial within 3 months prior to dosing.
* Investigator considered to be inappropriate for enrollment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Taneasy 600mg granules and Fluimucil 600MG granules administered twice daily for 14 days in treatment of COPD Disease. | one month
  Primary Evaluation Criteria:
  CAT score (COPD Assessment Test) The maximum score is 40. Higher scores indicate your COPD has a greater impact on your overall health and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No